CLINICAL TRIAL: NCT05527743
Title: Effectiveness of an Invasive Physical Therapy Protocol in Carpal Tunnel Syndrome: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFC22STC
Record Dates: First submitted 2022-08-26; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive Physiotherapy (Experimental)
  Interventions: Other: Invasive Physiotherapy
- Sham Group (Placebo Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: Invasive Physiotherapy — They will receive an invasive physiotherapy protocol of 3 sessions of percutaneous electrolysis and percutaneous neuromodulation guided by ultrasound, with a time margin of one week between the first and the second session and two weeks between the second and the third. Each session will last approximately 30 minutes. Each treatment session will consist of the application of 3 impacts of 3 seconds of 1.5mA intensity (1.5:3:3) (34), in a needle placed in an echoguided manner in the carpal tunnel in relation to the median nerve over the area of fibrosis or entrapment. Subsequently, a second needle will be placed ultrasound-guided at the level of the elbow crease in relation to the median nerve. A symmetric biphasic current with a frequency of 2Hz and a pulse width of 250µs (22,35) will be applied for 17 minutes (36), increasing the intensity of the current until a slight tolerable discomfort is produced in relation to the patient's symptomatology.
  Arms: Invasive Physiotherapy
Other: Sham — The participants of the study corresponding to the sham group will receive the application of the transcutaneous electrical stimulation sham technique (37), placing the patches in the same points where the needles are located in the percutaneous electrolysis and percutaneous neuromodulation technique, remaining in the supine position for the necessary time after the technique is performed, until 30 minutes are completed, thus ensuring that the evaluator does not know to which group each patient has been assigned (37). This technique has been studied as a sham technique for electrolysis and neuromodulation interventions (37).
  Once the study is completed and if the results are better in the IF group, the subjects in the sham group will be offered to receive this treatment. The reason for this is to ensure that the entire sample ends up receiving a treatment that, a priori, should improve their functional capacities, thus guaranteeing one of the ethical principles of research.
  Arms: Sham Group

SUMMARY:
Carpal Tunnel Syndrome (CTS) is the most common peripheral neuropathy due to entrapment, caused by compression of the median nerve as it passes under the transverse carpal ligament at the wrist. The prevalence of CTS is between 5% and 20% in the general population, according to the criteria used. It stands at 10% when following the criteria established by the National Institute for Occupational Safety and Health.

Within the prevalence, 1% are men and 7% women, with an incidence per year of 105 cases per 100,000 people. In 2019, the external consultant "statista" indicated that approximately 924,000 cases of CTS were registered in Spain. CTS generates large saturations in rehabilitation in primary care and in preoperative lists, for example, in 2008 there were 4,109 hospital admissions with a rate of 0.18 hospital discharges per thousand.

Risk factors for the development of CTS include female sex, older age, diabetes, menopause, hypothyroidism, obesity and pregnancy. Smoking appears to be a risk factor in the development of CTS. As well as wrist hyperflexion and hyperextension movements. The number of risk factors present progressively increases the prevalence of CTS.

CTS is characterized by the presence of neuropathic pain, nocturnal paresthesias and dysesthesia. It can be combined with loss of strength and atrophy of the tenar muscles. Therefore, the most severe cases produce very notable physical, psychological and economic consequences. For example, in the United States, CTS generates an annual primary care expenditure of $2 billion. Currently, the most recent clinical guidelines recommend the use of orthoses, exercises and manual therapy in the management of CTS, although there is no consensus on the most effective option. On the other hand, surgery is one of the most used therapeutic options. However, there is a great collapse of the health system and the waiting list for the intervention and it can take a long time.

The conservative therapeutic options used to date focus on the local approach to CTS at the wrist, and a recent systematic review has shown a high rate of surgical need (around 60%) at 3-year follow-up. This need for surgery may be reduced in the long term to 15% if the conservative approach includes maneuvers focused on desensitization of the central nervous system, performing an approach to the entire upper extremity. Current evidence suggests that CTS is a complex disorder, which presents sensitization mechanisms of the nervous system, and not only a peripheral nerve compression at the carpal tunnel level. Therefore, approaches and therapies with a central effect are hypothesized to be of future interest, in accordance with current nociceptive theories of CTS.

In the field of physiotherapy, novel techniques have been developed in recent years, such as ultrasound-guided percutaneous musculoskeletal electrolysis and ultrasound-guided percutaneous neuromodulation, in which different types of electrical current are applied through solid needles.

Different mechanisms of action have been associated with these invasive techniques, such as a potential effect on the activation of the descending pain inhibitory system pathways, the reduction of evoked motor potentials and an increase in intracortical inhibition, suggesting benefits in patients with central sensitization.

Invasive electrolysis and neuromodulation techniques have been applied in other studies at the nerve level, especially in the sciatic nerve at the piriformis and hamstrings level, in the popliteal fossa and in the foot. However, there is no study performed in patients with CTS.

To date, there is no clear consensus on the therapeutic approach to CTS, and the application of these invasive physiotherapy techniques is a novel approach that encompasses the local effect of treatment by means of local ultrasound-guided insertion of the needle in the carpal tunnel and the central neurophysiological effect produced by the current when it is applied. Taking into account the good empirical results found in private clinics and the precedents of studies carried out in other nerves, this treatment approach for outpatient application in primary care centers could relieve the demand for hospital care for patients referred for surgical treatment.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is the most common peripheral neuropathy due to entrapment, caused by compression of the median nerve as it passes under the transverse carpal ligament at the wrist. The prevalence of CTS is between 5% and 20% in the general population, according to the criteria used. It stands at 10% when following the criteria established by the National Institute for Occupational Safety and Health.

Within the prevalence, 1% are men and 7% women, with an incidence per year of 105 cases per 100,000 people. In 2019, the external consultant "statista" indicated that approximately 924,000 cases of CTS were registered in Spain. CTS generates large saturations in rehabilitation in primary care and in preoperative lists, for example, in 2008 there were 4,109 hospital admissions with a rate of 0.18 hospital discharges per thousand.

Risk factors for the development of CTS include female sex, older age, diabetes, menopause, hypothyroidism, obesity and pregnancy. Smoking appears to be a risk factor in the development of CTS. As well as wrist hyperflexion and hyperextension movements. The number of risk factors present progressively increases the prevalence of CTS.

CTS is characterized by the presence of neuropathic pain, nocturnal paresthesias and dysesthesia. It can be combined with loss of strength and atrophy of the tenar muscles. Therefore, the most severe cases produce very notable physical, psychological and economic consequences. For example, in the United States, CTS generates an annual primary care expenditure of $2 billion. Currently, the most recent clinical guidelines recommend the use of orthoses, exercises and manual therapy in the management of CTS, although there is no consensus on the most effective option. On the other hand, surgery is one of the most used therapeutic options. However, there is a great collapse of the health system and the waiting list for the intervention and it can take a long time.

The conservative therapeutic options used to date focus on the local approach to CTS at the wrist, and a recent systematic review has shown a high rate of surgical need (around 60%) at 3-year follow-up. This need for surgery may be reduced in the long term to 15% if the conservative approach includes maneuvers focused on desensitization of the central nervous system, performing an approach to the entire upper extremity. Current evidence suggests that CTS is a complex disorder, which presents sensitization mechanisms of the nervous system, and not only a peripheral nerve compression at the carpal tunnel level. Therefore, approaches and therapies with a central effect are hypothesized to be of future interest, in accordance with current nociceptive theories of CTS.

In the field of physiotherapy, novel techniques have been developed in recent years, such as ultrasound-guided percutaneous musculoskeletal electrolysis and ultrasound-guided percutaneous neuromodulation, in which different types of electrical current are applied through solid needles.

Different mechanisms of action have been associated with these invasive techniques, such as a potential effect on the activation of the descending pain inhibitory system pathways, the reduction of evoked motor potentials and an increase in intracortical inhibition, suggesting benefits in patients with central sensitization.

Invasive electrolysis and neuromodulation techniques have been applied in other studies at the nerve level, especially in the sciatic nerve at the piriformis and hamstrings level, in the popliteal fossa and in the foot. However, there is no study performed in patients with CTS.

To date, there is no clear consensus on the therapeutic approach to CTS, and the application of these invasive physiotherapy techniques is a novel approach that encompasses the local effect of treatment by means of local ultrasound-guided insertion of the needle in the carpal tunnel and the central neurophysiological effect produced by the current when it is applied. Taking into account the good empirical results found in private clinics and the precedents of studies carried out in other nerves, this treatment approach for outpatient application in primary care centers could relieve the demand for hospital care for patients referred for surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or superior to 18 years old.
* Have a medical diagnosis of CTS, by a specialist of the Neurophysiology Service with confirmation of neurophysiological study, in any of its stages: mild, moderate or severe.
* Have access and be able (or have help) to use an online platform to conduct "meetings" with the health professional.
* Read the informed consent form and understand the objectives and conduct of the study.

Exclusion Criteria:

* Be pending compensation or litigation for health problems.
* Receiving physiotherapy treatment in the region in the month prior to the study.
* Present severe diseases that may be related to the clinical results: malignancy or history of cancer, tumors or fractures in the region to be treated, blood dyscrasia, severe trauma in the previous 3 months, surgery in the region in the previous 12 months.
* To present contraindications to the therapeutic approach such as Belanophobia (33).
* Subjects who have received any of the procedures under study (percutaneous neuromodulation or percutaneous electrolysis technique).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Present Pain Intensity (NPRS 0-10) | Baseline; 1 month follow-up; 6 month follow-up
  The intensity of hand pain will be recorded, using an 11-point numerical scale (NPRS) (0=no pain, 10=maximum pain). They will be asked for current pain. Because there is no value that determines the minimum clinically relevant difference in hand pain, a 2-point change, or 30% change, will be considered clinically relevant (38).
Change in Pain Intensity in the previous week (NPRS 0-10) | Baseline; 1 month follow-up; 6 month follow-up
  The intensity of hand pain will be recorded, using an 11-point numerical scale (NPRS) (0=no pain, 10=maximum pain). They will be asked for the worst pain experienced in the previous week. Because there is no value that determines the minimum clinically relevant difference in hand pain, a 2-point change, or 30% change, will be considered clinically relevant (38).

SECONDARY OUTCOMES:
Change in Neurophysiological study (m/s) | Baseline; 1 month follow-up; 6 month follow-up
  The procedures will be performed by a neurophysiologist with more than 10 years of clinical and research experience. The electrophysiological diagnostic criteria for CTS of the American Association of Neuromuscular and Electrodiagnostic Medicine (39) and the normal ranges of motor and sensory nerve conduction as described in the literature (40) will be used.
  The degree of electrophysiological compromise present will be classified according to the Bland scale (41). The following will be taken as study variables: existence of denervation, distal motor latency of median nerve and ulnar nerve, distal sensory latency of median nerve and ulnar nerve, conduction velocity, action potential amplitude and sensory detail of both.
Change in BOSTON questionnaire | Baseline; 1 month follow-up; 6 month follow-up
  Self-administered questionnaire designed to record symptom severity and functional status of patients with CTS (42). Higher scores are indicative of worse functional capacity and greater symptom severity. Minimally relevant clinical changes have been determined as 0.74 points for the function subscale and 1.14 points for the symptom severity subscale (43).
Change in Global rating of change scale | Baseline; 1 month follow-up; 6 month follow-up
  Scale of global change perceived by the patient, designed to detect improvement or deterioration of the patient over time (44). An 11-point numerical scale (-7=evolving to much worse; +7=fully recovered). Considering +4 and +5 moderate positive changes and +6 and +7 notable changes (45).
Change in Katz Diagram | Baseline; 1 month follow-up; 6 month follow-up
  Diagram for the localization of symptoms in the dorsal and palmar part of the hand, self-administered. The patient determines the location of his symptoms, determining them as pain, numbness, sensation of passing current or other. The diagnosis is considered as classic, probable, possible, or unlikely, according to Calfee (46).
Change in Grip strength (Newtons) | Baseline; 1 month follow-up; 6 month follow-up
  A single measurement of grip strength will be performed, which has been shown to be more reliable than the average of 3 attempts (47), with the dynamometer (Baseline 12-0241 LITE) in Newtons. The patient will be seated with shoulder and wrist in neutral position and elbow at 90º of flexion (48).
Change in Sensitivity (discrimination of two points) | Baseline; 1 month follow-up; 6 month follow-up
  The discrimination of two points on the palmar side of the 3rd target will be assessed, taking 6mm of distance as the normative value of discrimination of 2 points. Pressure will be applied with one or two points until causing some discomfort to the patient, having to discriminate if stimulated with 1 or 2 points, the minimum distance that manages to discriminate will be recorded (49).
Change in Sensitivity (Semmes-Weinstein Monofilament Test) | Baseline; 1 month follow-up; 6 month follow-up
  Stimulation by means of pressure filaments, seeking to detect the sensitive threshold by means of 1 second pressures, the necessary pressure will be applied to cause a slight deformation of the filament. The lightest filament detected (50) will be recorded.
Change in Inhibitory modulation conditioned by pain (Kpa) | Baseline; 1 month follow-up; 6 month follow-up
  It will be performed with the aim of exploring the descending inhibitory pathway (51). The test of pain thresholds by pressure in the affected area is performed. A remote area, usually arm or hand, is subjected to a painful stimulus (ice cube) (52) or ischemia cuff (maximum 10 min at 200 mmHg or up to VAS 6). At that time, the pressure pain threshold test is repeated on the affected area. An increase in the value of the pressure threshold test will denote a correct functioning of the inhibitory modulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Derived] Borrella-Andres S, Rodriguez-Sanz J, Lopez-de-Celis C, Marques Garcia I, Bueno-Gracia E, Rodriguez-Mena D, Malo-Urries M. Effect of ultrasound-guided percutaneous electrolysis and nerve stimulation on pain and function in carpal tunnel syndrome: A randomized clinical trial. Pain Med. 2025 Dec 4:pnaf170. doi: 10.1093/pm/pnaf170. Online ahead of print. PMID 41528761